CLINICAL TRIAL: NCT07117669
Title: A Phase 1/2, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation and Expansion Study of ENP-501 in Non-Peanut Allergic Participants and Participants With a Known Peanut Allergy
Brief Title: Study of ENP-501 in Peanut-Allergic and Non-Allergic Participants
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: N-Fold, LLC (Industry)
Collaborators: CBCC Global Research (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENP-501-001
Record Dates: First submitted 2025-08-04; First posted 2025-08-12 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Peanut Allergy
Keywords: Peanut Hypersensitivity
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ENP-501 (Experimental)
  Interventions: Drug: ENP-501
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ENP-501 — * Part 1: Participants will receive buccal administrations of ENP-501 daily for 6-14 weeks
  * Part 2: Participants will receive buccal administrations of ENP-501 daily for 52 weeks following achieving the 2000 µg target dose
  Arms: ENP-501
Drug: Placebo — * Part 1: Participants will receive buccal administrations of placebo daily for 6-14 weeks
  * Part 2: Participants will receive buccal administrations of placebo daily for 52 weeks following achieving the 2000 µg target dose
  Arms: Placebo

SUMMARY:
This is a Phase 1/2 study to evaluate the safety and clinical activity of ENP-501 in non-peanut allergic (NPA) healthy participants and participants with an established peanut allergy (PA)

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* 14-50 years of age (inclusive)
* Otherwise medically healthy and able to participate in the study
* Able to perform spirometry testing in accordance with the American Thoracic Society (ATS) guidelines (2019)
* All women of child-bearing potential, agree to either abstain from sexual activity or agree to use an adequate method of contraception for the duration of the study and for 30 days after the last dose of investigational product
* Signed and dated written informed consent from the participant and/or parent or guardian
* Signed and dated assent from participant under 18 in accordance with local IRB regulations
* Willing and able to avoid peanut and peanut contaminants for the duration of the trial

Part 1 Cohort 1 only (NPA Participants)

* No known clinical history of peanut allergy with regular exposure to peanuts in daily life, i.e ingests peanuts without symptoms
* Negative Skin Prick Test (SPT) (wheal diameter of <3 mm) to peanut

Part 1 Cohort 2 only (PA Participants)

* A documented clinical history of peanut allergy, which includes the development of symptoms (e.g., urticaria, flushing, rhinorrhea and sneezing, throat tightness or hoarseness, wheezing, vomiting) verified by a physician
* At least two of the three following requirements:

  1. Positive Skin Prick Test (SPT) (wheal diameter of ≥ 8 mm) to peanut
  2. An elevated serum peanut specific IgE level ≥ 7 kUA/L (ImmunoCAP®)
  3. An Ara-h2 IgE level of ≥ 2 kUA/L (ImmunoCAP®)

Part 2:

* 14 to 50 years of age (inclusive)
* A documented clinical history of peanut allergy, which includes the development of symptoms (e.g., urticaria, flushing, rhinorrhea and sneezing, throat tightness or hoarseness, wheezing, vomiting) verified by a physician
* At least two of the three following requirements at screening:

  1. Positive SPT (wheal diameter of ≥ 3 mm) to peanut
  2. Serum peanut-specific IgE level ≥ 0.7 kUA/L (ImmunoCAP®)
  3. An Ara-h2 IgE level of ≥ 0.5 kUA/L (ImmunoCAP®) within 1 year of enrollment
* Participant must be willing and able to complete a DBPCFC at screening and EOT (24-hours after last dose) and experience dose-limiting symptoms at or before the 300 mg challenge dose of peanut protein during a Double Blind, Placebo Controlled Food Challenge (DBPCFC) conducted in accordance with Practical Issues in Allergology, Joint United States/European Union Initiative (PRACTALL) guidelines
* Otherwise medically healthy and able to participate in the study
* Able to perform spirometry testing in accordance with the ATS guidelines (2019)
* All women of child-bearing potential, agree to either abstain from sexual activity or agree to use an adequate method of contraception for the duration of the study and for 30 days after the last dose of investigational product
* Signed and dated written informed consent from the participant and/or parent or guardian
* Signed and dated assent from participant under 18 in accordance with local IRB regulations
* Willing and able to avoid peanut and peanut contaminants for the duration of the trial

Exclusion Criteria:

* History of severe anaphylactic event requiring mechanical ventilation or use of intravenous (IV) vasopressor drugs
* Clinically significant screening electrocardiogram (ECG) abnormality or corrected QTcF >/= 450 msec at Screening
* FEV1 value < 80% predicted at Screening
* Any hospitalization in the past year for asthma, >1 course of oral steroids for asthma in the past 6 months, or any emergency room visit in the past 6 months for asthma
* Poorly controlled atopic dermatitis
* Eosinophilic gastrointestinal disease
* Use of oral or IV corticosteroids within 30 days of Screening
* Use of tricyclic antidepressants within 6 months of Screening
* Inability to discontinue antihistamines for at least 5 half-lives before skin testing
* Use of omalizumab or other immunomodulatory therapy (not including corticosteroids) or biologic therapy within one year of Screening
* Use of any food allergen-specific or other non-traditional form of allergen immunotherapy within one year of Screening
* Use of immunosuppressive drugs within 30 days of Screening
* Use of ß-blockers (oral)
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urinalysis
* Pregnant or breast-feeding (if female)
* Behavioral, cognitive, or psychiatric disease that in the opinion of the Investigator affects the ability of the participant to understand and cooperate with the study protocol
* Known allergy to inactive ingredients of investigational product (active or placebo)
* Participation in another interventional clinical trial within 30 days of Screening or within 5 half-lives of the other IP
* Residing at the same address as another participant in this or any peanut immunotherapy study

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) as Assessed by NCI CTCAE v 5.0 in Part 1 | Up to 22 Weeks
Number of Participants with Treatment-Emergent Serious Adverse Events (TESAEs) as Assessed by NCI CTCAE v 5.0 in Part 1 | Up to 22 Weeks
Number of Participants with Dose Limiting Toxicities (DLTs) as Assessed by NCI CTCAE v 5.0 in Part 1 | Up to 22 Weeks
Number of Participants with Systemic Reactions as Assessed by NCI CTCAE v 5.0 in Part 1 | Up to 22 Weeks
Number of Participants with changes in Clinical Laboratory Values in Part 1 | Up to 22 Weeks
Number of Participants with changes in Physical Examination in Part 1 | Up to 22 Weeks
Number of Participants with changes in Vital Signs in Part 1 | Up to 22 Weeks
Proportion of Participants Tolerating ≥1043 mg Cumulative Peanut Protein Without Dose-Limiting Symptoms at End of Treatment (EOT) Visit Double-Blind Placebo-Controlled Food Challenge (DBPCFC) Compared to Placebo in Part 2 | Up to 72 Weeks

SECONDARY OUTCOMES:
Number of Participants Able to Tolerate 2000 µg Dose of ENP-501 Without Experiencing Dose-Limiting Toxicity (DLT) in Part 1 | Up to 22 Weeks
Change in Total IgE Levels in Part 1 | Screening and Week 22 (EOS)
Change in Ara h 1-Specific IgE Levels in Part 1 | Screening and Week 22 (EOS)
Change in Ara h 2-Specific IgE Levels in Part 1 | Screening and Week 22 (EOS)
Change in Ara h 3-Specific IgE Levels in Part 1 | Screening and Week 22 (EOS)
Change in Ara h 1-Specific IgG4 Levels in Part 1 | Screening and Week 22 (EOS)
Change in Ara h 2-Specific IgG4 Levels in Part 1 | Screening and Week 22 (EOS)
Change in Ara h 3-Specific IgG4 Levels in Part 1 | Screening and Week 22 (EOS)
Change in Wheal Diameter on Skin Prick Test (SPT) to Peanut in Part 1 | Screening and Week 22 (EOS)
Proportion of Participants Tolerating at Least 443 mg Cumulative Dose of Peanut Protein Without Dose-Limiting Symptoms at EOT Visit DBPCFC Compared to Placebo in Part 2 | Up to 72 Weeks
Proportion of Participants Tolerating at Least 2043 mg Cumulative Dose of Peanut Protein Without Dose-Limiting Symptoms at EOT Visit DBPCFC Compared to Placebo in Part 2 | Up to 72 Weeks
Proportion of Participants Tolerating 4043 mg Cumulative Dose of Peanut Protein Without Dose-Limiting Symptoms at EOT Visit DBPCFC Compared to Placebo in Part 2 | Up to 72 Weeks
Maximum Severity of Symptoms Occurring at Each Challenge Dose of Peanut Protein During the Exit DBPCFC in Part 2 | Up to 72 Weeks
Number of Participants Able to Tolerate the 2000 µg Dose of ENP-501 in Part 2 | Up to 72 Weeks
Change in Total IgE Levels in Part 2 | Screening and Week 72 (EOS)
Change in Ara h 1-Specific IgE Levels in Part 2 | Screening and Week 72 (EOS)
Change in Ara h 2-Specific IgE Levels in Part 2 | Screening and Week 72 (EOS)
Change in Ara h 3-Specific IgE Levels in Part 2 | Screening and Week 72 (EOS)
Change in Ara h 1-Specific IgG4 Levels in Part 2 | Screening and Week 72 (EOS)
Change in Ara h 2-Specific IgG4 Levels in Part 2 | Screening and Week 72 (EOS)
Change in Ara h 3-Specific IgG4 Levels in Part 2 | Screening and Week 72 (EOS)
Change in Wheal Diameter on Skin Prick Test (SPT) to Peanut in Part 2 | Screening and Week 72 (EOS)
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) as Assessed by NCI CTCAE v 5.0 in Part 2 | Up to 72 Weeks
Number of Participants with Treatment-Emergent Serious Adverse Events (TESAEs) as Assessed by NCI CTCAE v 5.0 in Part 2 | Up to 72 Weeks
Number of Participants with TEAEs leading to discontinuation as Assessed by NCI CTCAE v 5.0 in Part 2 | Up to 72 Weeks
Number of Participants with Systemic Reactions as Assessed by NCI CTCAE v 5.0 in Part 2 | Up to 72 Weeks
Number of Participants with changes in Clinical Laboratory Values in Part 2 | Up to 72 Weeks
Number of Participants with changes in Physical Examination in Part 2 | Up to 72 Weeks
Number of Participants with changes in Vital Signs in Part 2 | Up to 72 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site 001, Aurora, Colorado, United States